CLINICAL TRIAL: NCT02570295
Title: Swiss Army Physical Fitness Training - An Intervention Study Investigating the Influence of the Swiss Armed Forces' New Sport Concept on Physical and Psychological Parameters of the Recruits
Brief Title: Swiss Army Physical Fitness Training
Acronym: SAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Sport Magglingen (Other Government)
Collaborators: Swiss Armed Forces (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAFT_82/15
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Wounds and Injuries; Physical Activity; Mood (Psychological Function); Motivation; Motor Activity
Keywords: Army; Sport; Physical Fitness; Injuries; Psychological Tests; Attrition
MeSH Terms: conditions — Wounds and Injuries; Motor Activity; Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swiss Army Physical Fitness Training (Experimental): Sport according to the new sport concept ("Swiss Army Physical Fitness Training") of the Swiss Armed Forces
  Interventions: Other: Swiss Army Physical Fitness Training
- Traditional Sport Concept (No Intervention): Sport according to the traditional sport concept of the Swiss Armed Forces

INTERVENTIONS:
Other: Swiss Army Physical Fitness Training — 2 x 90 minutes strength training and sport games and 2 x 30 minutes endurance training per week during 18 weeks of basic military training
  Arms: Swiss Army Physical Fitness Training

SUMMARY:
The purpose of this study is to determine whether the new sport concept of the Swiss Armed Forces influences the physical and psychological fitness of the recruits.

DETAILED DESCRIPTION:
The physical and psychological demands in the Swiss Army basic military service are high. Injury incidences in Swiss Army training schools are higher than in armed forces of other countries.There is evidence that progressive loading of physical demands at the beginning of basic military service and specific physical training can reduce injury incidences and attrition rates. A new sport concept by the Swiss Army takes into account these results of previous studies. Therefore, the aim of this study is to investigate the influences of this new sport concept on the physical and psychological fitness as well as on the injury and attrition rates of the recruits.

ELIGIBILITY:
Inclusion Criteria:

* Recruits of the Swiss Army rescue training schools 75 2/2015 and 3/2015

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 722 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wyss, PhD, Principal Investigator — Swiss Federal Institute of Sport Magglingen
Locations (1):
- Casern of the Swiss Army rescue training school 75, Wangen an der Aare, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roos L, Boesch M, Sefidan S, Frey F, Mader U, Annen H, Wyss T. Adapted marching distances and physical training decrease recruits' injuries and attrition. Mil Med. 2015 Mar;180(3):329-36. doi: 10.7205/MILMED-D-14-00184. PMID 25735025
- [Background] Wyss T, Roos L, Hofstetter MC, Frey F, Mader U. Impact of training patterns on injury incidences in 12 Swiss Army basic military training schools. Mil Med. 2014 Jan;179(1):49-55. doi: 10.7205/MILMED-D-13-00289. PMID 24402985
- [Background] Hofstetter MC, Mader U, Wyss T. Effects of a 7-week outdoor circuit training program on Swiss Army recruits. J Strength Cond Res. 2012 Dec;26(12):3418-25. doi: 10.1519/JSC.0b013e318245bebe. PMID 22190160
- [Background] Wyss T, Mader U. Energy expenditure estimation during daily military routine with body-fixed sensors. Mil Med. 2011 May;176(5):494-9. doi: 10.7205/milmed-d-10-00376. PMID 21634292
- [Background] Wyss T, Mader U. Recognition of military-specific physical activities with body-fixed sensors. Mil Med. 2010 Nov;175(11):858-64. doi: 10.7205/milmed-d-10-00023. PMID 21121495
- [Background] Wyss, T, Marti, B, Rossi, S, Kohler, U, & Mäder, U (2007). Assembling and Verfification of a Fitness Test Battery for the Recruitment of the Swiss Army and Nation-wide Use. Schweizerische Zeitschrift für
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Schumacher, J, Leppert, K, Gunzelmann, T, Strauss, B, & Brähler, E(2005). Die Resilienzskala - Ein Fragebogen zur Erfassung der psychischen Widerstandsfähigkeit als Personmerkmal. Zeitschrift für klinische Psychologie, Psychiatrie und Psychotherapie, 53(1), 16-39.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Started | 375 | 347
Completed | 364 | 289
Not Completed | 11 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept | Total
Number analyzed (Participants) | 375 | 347 | 722
Age, Customized [Number; unit: participants]
  18-25 years | 375 | 347 | 722
Sex/Gender, Customized [Number; unit: participants]
  male | 375 | 347 | 722

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Injuries
Description: All injuries which are registered in the patient's medical record are collected and classified. A classification system which takes into account anatomical site, circumstances of the accident, and severity of the injury is used.
Time Frame: During the basic military training (18 weeks)
Population: The overall number of participants analyzed is smaller than the corresponding numbers in the participant flow module, because only participants who finished the whole 18-weeks basic military training were included in the analysis.
Measure: Number; unit: participants with injuries
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 278 | 262
participants with injuries | 184 | 172

2. Secondary Outcome: Physical Fitness Measured With the Swiss Physical Fitness Test Battery (SPFTB)
Description: Physical Fitness is measured with the Swiss physical fitness test battery (SPFTB).
  The SPFTB contains a progressive endurance run, a trunk muscle strength test, a standing long jump, a seated shot put, and a one-leg standing test. From the results of those performance tests (0 to 25 points each), a total fitness score is calculated (sum of all points). The minimum total score (worst result) is 0 points, the maximum total score (best result) is 125 points. A detailed description of the SPFTB can be found in the publication of Wyss, Marti, Rossi, Kohler and Mäder (2007).
Time Frame: Weeks 2, 10 and 16 of the basic military training
Population: The overall number of participants analyzed is smaller than the corresponding number in the participant flow module, because only participants who completed all three fitness tests were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 125
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 97 | 109
units on a scale from 0 to 125
  fitness test week 2 | 73.54 (12.83) | 73.56 (11.55)
  fitness test week 10 | 81.78 (11.27) | 77.16 (10.85)
  fitness test week 16 | 72.84 (13.43) | 65.05 (12.29)

3. Secondary Outcome: Psychological Questionnaires
Description: 2 questionaires concerning resilience were used: The Resilience Scale 11 (Schumacher, Leppert, Gunzelmann, Strauss & Brähler, 2005) and the Brief Resilience Scale (Smith, Dalen, Wiggings, Tooley, Christopher & Bernard, 2008). A mean was calculated for each time point. The total score ranges from 1 (worst result) to 7 (best result).
Time Frame: Weeks 2, 10 and 16 of the basic military training
Population: The overall number of participants analyzed is smaller than the corresponding number in the participant flow module, because only participants who the psychological questionnaires at all three time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale 1-7
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 23 | 29
units on a scale 1-7
  Resilience week 2 | 4.96 (1.09) | 5.14 (0.75)
  Resilience week 10 | 5.24 (1.05) | 5.46 (0.80)
  Resilience week 16 | 5.36 (0.85) | 5.48 (0.82)

4. Secondary Outcome: Military Performance According to Military Marks
Description: Military marks are given by superior Army personnel. The total score ranges from 1 (insufficient) to 5 (excellent). In total, three marks are given during the whole basic military training (after 7, 11 and 16 weeks). Data from those three time points are combined in a single value (mean).
Time Frame: During the basic military training (18 weeks)
Population: The overall number of participants analyzed is smaller than the corresponding number in the participant flow module, because only participants from whom military marks were available for the whole basic military training were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale 1-5
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 187 | 203
units on a scale 1-5 | 3.06 (0.37) | 2.91 (0.31)

5. Secondary Outcome: Questionnaire About Health and Physical Activities
Time Frame: Week 1 of the basic military training and 3 months after finishing the basic military training
Population: The overall number of participants analyzed is smaller than the corresponding number in the participant flow module, because only participants who completed the questionnaire at both time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: Minutes of physical activity per week
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 54 | 48
Minutes of physical activity per week
  Week 1 of basic military training | 969.19 (1171.67) | 717.69 (936.98)
  3 months after basic military training | 1251.37 (2297.40) | 845.02 (1088.230)

6. Secondary Outcome: Attrition Rate
Description: Withdrawals from the military service are reported by the training school's secretariat
Time Frame: During the whole basic military training (18 weeks)
Measure: Number; unit: participants
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 375 | 347
participants | 45 | 41

7. Other Pre Specified Outcome: Questionnaire About Sport Lessons
Description: Duration of each sport session was registered in a questionnaire by the military personnel. The minimum would be 0 minutes of sport per week, for the maximum the scale is open-ended. Data of sport lessons during the whole basic military are combined and presented as a mean value for each group.
Time Frame: During the whole basic military training (18 weeks)
Measure: Mean (Standard Deviation); unit: minutes of sport per week
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 375 | 347
minutes of sport per week | 182.53 (62.72) | 113.17 (72.7)

8. Other Pre Specified Outcome: Daily Energy Expenditure
Description: Daily energy expenditure was measured using two accelerometers and one heart rate sensor. Data from weeks 2-9 of the basic military were combined and a single value (mean) was calculated for each group.
Time Frame: Weeks 2 - 9 of the basic military training
Population: The overall number of participants analyzed is smaller than the corresponding number in the participant flow module, because only an exemplary sample of 40 participants per group were chosen to wear the sensors due to financial reasons.
Measure: Mean (Standard Deviation); unit: Megajoule per day
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 40 | 40
Megajoule per day | 12.02 (0.65) | 10.45 (0.84)

9. Other Pre Specified Outcome: Daily Distance Covered on Foot
Description: Daily distance covered on foot was measured using two accelerometers and one heart rate sensor. Data from weeks 2-9 of the basic military were combined and a single value (mean) was calculated for each group.
Time Frame: Weeks 2 - 9 of the basic military training
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: km per day
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Number analyzed (Participants) | 40 | 40
km per day | 15.66 (1.77) | 14.22 (1.86)

ADVERSE EVENTS:
Arm/Group | Swiss Army Physical Fitness Training | Traditional Sport Concept
Serious Adverse Events (participants affected / at risk) | 0/375 | 0/347
Other Adverse Events (participants affected / at risk) | 0/375 | 0/347

LIMITATIONS AND CAVEATS:
It is possible that people who are interested in health or fitness issues were more likely to sign the informed consent, which could have had an influence on the injuries and fitness outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes